CLINICAL TRIAL: NCT03172182
Title: The Effects of Operating Room Virtual Tour on Preoperative Anxiety, Emergence Delirium and Postoperative Behavioral Changes of Pediatric Patients: Prospective, Randomized, and Controlled Trial
Brief Title: Perioperative Effects of Operating Room Virtual Tour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sung-Hee Han, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-1705-396-302
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Preoperative Care; Anxiety; Emergence Delirium; Postoperative Complications
MeSH Terms: conditions — Anxiety Disorders; Emergence Delirium; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (VR) group (Experimental): Immersive education using a 360-degree VR video tour at operation day
  Interventions: Behavioral: a 360-degree VR video tour
- Control Group (No Intervention): Conventional verbal education of preoperative proceudres

INTERVENTIONS:
Behavioral: a 360-degree VR video tour — At operation day, pediatric patients of the VR group and their parents are educated using virtual tour program explaining preoperative procedures and showing environment of the operating room. A 360-degree virtual reality (VR) video for the tour program was filmed in advance and is provided using a head mount device into which a smartphone is installed, at 30 minutes before the induction of anesthesia.
  Arms: Virtual reality (VR) group

SUMMARY:
Preoperative anxiety is associated with adverse consequences such as emergence delirium, and postoperative behavioral changes. According to previous studies, providing information of anesthetic procedures helps to lessen preoperative anxiety. However, verbal explanation alone provides the limited effect, and the tour program of the operating room prior to surgery may not be possible for a number of hospitals due to organizational and financial reasons. Therefore, the virtual reality (VR) tour of the operating room may be an innovative and novel method to give children information about the preoperative process and to alleviate the preoperative anxiety. In this study, we intend to evaluate the effects of the operating room virtual tour on preoperative anxiety as well as emergence delirium and postoperative behavioral changes, in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* American Society of Anesthesiologist (ASA) physical class I, II
* Informed consent; Children aged between 4 and 6 years old are allowed to have verbal consent and their parents provide informed written consent. Children over the age of 7 are required to obtain a written consent with parental permission.

Exclusion Criteria:

* ASA class ≥ III
* Major surgery needing postoperative intensive care unit (ICU) admission.
* Chronic disease or history of preterm birth
* Developmental delay
* Hearing or vision impairment
* Affective disorder
* History of epilepsy or seizure
* Previous experience of general anesthesia

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Emergence delirium | At 5 minutes after arrival in post-anesthesia care unit (PACU)
  Pediatric Anesthesia Emergence Delirium (PAED) scale

SECONDARY OUTCOMES:
Preoperative anxiety | 2 times; before the intervention (baseline) and, at waiting area, before the operating room entrance (preoperative)
  Modified Yale Preoperative Anxiety Scale (mYPAS)
Postoperative behavioral change | 2 times; on the 1st and 14th day (2 weeks) after the surgery, we will call and talk with the parents
  Hospitalization Post- Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hee Han, MD/PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moura LA, Dias IM, Pereira LV. Prevalence and factors associated with preoperative anxiety in children aged 5-12 years. Rev Lat Am Enfermagem. 2016 Jun 14;24:e2708. doi: 10.1590/1518-8345.0723.2708. PMID 27305179
- [Background] Wollin SR, Plummer JL, Owen H, Hawkins RM, Materazzo F. Predictors of preoperative anxiety in children. Anaesth Intensive Care. 2003 Feb;31(1):69-74. doi: 10.1177/0310057X0303100114. PMID 12635399
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Thompson RH, Vernon DT. Research on children's behavior after hospitalization: a review and synthesis. J Dev Behav Pediatr. 1993 Feb;14(1):28-35. PMID 8432876
- [Background] Chrousos GP, Gold PW. The concepts of stress and stress system disorders. Overview of physical and behavioral homeostasis. JAMA. 1992 Mar 4;267(9):1244-52. PMID 1538563
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Background] Arai YC, Ito H, Kandatsu N, Kurokawa S, Kinugasa S, Komatsu T. Parental presence during induction enhances the effect of oral midazolam on emergence behavior of children undergoing general anesthesia. Acta Anaesthesiol Scand. 2007 Aug;51(7):858-61. doi: 10.1111/j.1399-6576.2007.01339.x. Epub 2007 Jun 18. PMID 17578463
- [Background] El Batawi HY. Effect of preoperative oral midazolam sedation on separation anxiety and emergence delirium among children undergoing dental treatment under general anesthesia. J Int Soc Prev Community Dent. 2015 Mar-Apr;5(2):88-94. doi: 10.4103/2231-0762.155728. PMID 25992332
- [Background] Rice M, Glasper A, Keeton D, Spargo P. The effect of a preoperative education programme on perioperative anxiety in children: an observational study. Paediatr Anaesth. 2008 May;18(5):426-30. doi: 10.1111/j.1460-9592.2008.02490.x. PMID 18384339
- [Background] Sadegh Tabrizi J, Seyedhejazi M, Fakhari A, Ghadimi F, Hamidi M, Taghizadieh N. Preoperative Education and Decreasing Preoperative Anxiety Among Children Aged 8 - 10 Years Old and Their Mothers. Anesth Pain Med. 2015 Aug 22;5(4):e25036. doi: 10.5812/aapm.25036. eCollection 2015 Aug. PMID 26473103
- [Background] Kerimoglu B, Neuman A, Paul J, Stefanov DG, Twersky R. Anesthesia induction using video glasses as a distraction tool for the management of preoperative anxiety in children. Anesth Analg. 2013 Dec;117(6):1373-9. doi: 10.1213/ANE.0b013e3182a8c18f. PMID 24257388
- [Background] Liguori S, Stacchini M, Ciofi D, Olivini N, Bisogni S, Festini F. Effectiveness of an App for Reducing Preoperative Anxiety in Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):e160533. doi: 10.1001/jamapediatrics.2016.0533. Epub 2016 Aug 1. PMID 27294708
- [Background] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Background] Makkar JK, Bhatia N, Bala I, Dwivedi D, Singh PM. A comparison of single dose dexmedetomidine with propofol for the prevention of emergence delirium after desflurane anaesthesia in children. Anaesthesia. 2016 Jan;71(1):50-7. doi: 10.1111/anae.13230. Epub 2015 Oct 7. PMID 26444149
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Jenkins BN, Kain ZN, Kaplan SH, Stevenson RS, Mayes LC, Guadarrama J, Fortier MA. Revisiting a measure of child postoperative recovery: development of the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery. Paediatr Anaesth. 2015 Jul;25(7):738-45. doi: 10.1111/pan.12678. Epub 2015 May 9. PMID 25958978

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03172182/Prot_SAP_000.pdf